CLINICAL TRIAL: NCT04162691
Title: Single Cell Sequencing Analysis of Thymoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, ZHAO An, Principal Investigator, Zhejiang Cancer Hospital
Other Study IDs: SCS-001
Record Dates: First submitted 2019-11-06; First posted 2019-11-14 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Thymoma
MeSH Terms: conditions — Thymoma | interventions — Histocompatibility Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Malignant thymoma
  Interventions: Diagnostic Test: Tissue
- Benign thymoma
  Interventions: Diagnostic Test: Tissue

INTERVENTIONS:
Diagnostic Test: Tissue — Four 4-5 mm tissues of the thymoma

SUMMARY:
The purpose of this study is to understand how genetics play a role in thymoma. Intratumoral heterogeneity is among the greatest challenges in precision cancer therapy. However, developments in high-throughput single-cell RNA sequencing (scRNA-seq) may now provide the statistical power to dissect the diverse cellular populations of tumors. This study aims to find out how it affects genetic and protein expression in patients with malignant thymoma, compared to Benign thymoma, at a single-cell level using a flow cytometry and RNA-sequencing protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with thymoma
* Ability to provide written consent and comply with the protocol
* At least 18 years of age

Exclusion Criteria:

* Patients undergoing thymoma treatment
* Patients with previous malignancy
* Known HIV positive status.
* Evidence of abnormality of any immune cell population from a drug-induced or genetic cause.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred to the clinic for investigation of a suspected thymoma condition
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-06-06 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Determination of cell population from thymoma | through study completion, an average of 1 year
  The genes expression and the cell population

CONTACTS AND LOCATIONS:
Locations (1):
- An Zhao, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers